CLINICAL TRIAL: NCT00461708
Title: An Open Label Study of Tarceva in Combination With Gemcitabine in Unresectable and/or Metastatic Cancer of the Pancreas : Relationship Between Skin Rash and Survival
Brief Title: A Study of Tarceva (Erlotinib) in Combination With Gemcitabine in Unresectable and/or Metastatic Cancer of the Pancreas: Relationship Between Skin Toxicity and Survival
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20296
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

ARMS (2):
- Rash, Grade <2 (Experimental): Participants with a rash graded less than (<) 2 according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version (v.) 3.0 received erlotinib, 100 milligrams (mg), orally (PO), once per day until disease progression, unacceptable toxicity or refusal of patient to continue with the treatment. Participants also received gemcitabine, 1000 mg per (/) square meter (m^2), intravenously (IV), over 30 minutes on Days 1, 8 and 15 in 4-week cycles until disease progression, unacceptable toxicity or refusal of patient to continue with the treatment.
  Interventions: Drug: Erlotinib; Drug: Gemcitabine
- Rash, Grade ≥2 (Experimental): Participants with a rash graded greater than or equal to (≥) 2 according to the NCI-CTC v. 3.0 received erlotinib, 100 mg, PO, once per day until disease progression, unacceptable toxicity or refusal of patient to continue with the treatment. Participants also received gemcitabine, 1000 mg/m^2, IV, over 30 minutes on Days 1, 8 and 15 in 4-week cycles until disease progression, unacceptable toxicity or refusal of patient to continue with the treatment.
  Interventions: Drug: Erlotinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Erlotinib — 100 mg, PO, once per day
  Other Names: Tarceva
Drug: Gemcitabine — 1000 mg/m2, IV, on Days 1, 8 and 15 in 4-week cycles

SUMMARY:
This single arm study will evaluate the relationship between the skin toxicity of Tarceva in combination with gemcitabine, and survival, in patients with advanced and/or metastatic pancreatic cancer. All patients will receive gemcitabine 100mg/m2 i.v. weekly; Tarceva will be administered 100mg po per day. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* locally advanced and/or metastatic pancreatic cancer (stage III or IV);
* Karnofsky performance Status of >=60%.

Exclusion Criteria:

* local(stage IA to IIB) pancreatic cancer;
* <=6 months since last adjuvant chemotherapy;
* previous systemic therapy for metastatic pancreatic cancer;
* other primary tumor within last 5 years (except for adequately treated cancer in situ of cervix, or basal cell skin cancer);
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Spain (24):
  - Alcoy, Alicante
  - Elche, Alicante
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Manresa, Barcelona
  - Sabadell, Barcelona, Barcelona
  - Santander, Cantabria
  - Córdoba, Cordoba
  - Girona, Girona
  - Granada, Granada
  - Guadalajara, Guadalajara
  - Jaén, Jaen
  - A Coruña, La Coruña
  - Lleida, Lerida
  - Lugo, Lugo
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Murcia, Murcia
  - Navarra, Navarre
  - Pontevedra, Pontevedra
  - Seville, Sevilla
  - Sagunto, Valencia
  - Valencia, Valencia
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib, Gemcitabine: Rash Grade Less Than (<) 2: Participants with a rash Grade < 2 according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version (V) 3.0 received erlotinib, 100 milligrams (mg), orally (PO), once per day of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant. Participants also received gemcitabine, 1000 milligrams per square meter (mg/m^2), intravenously (IV), over 30 minutes on Days 1, 8 and 15 of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant.
- Erlotinib, Gemcitabine: Rash Grade Greater Than/Equal to (≥) 2: Participants with a rash Grade ≥ 2 according to the NCI-CTC V 3.0 received erlotinib, 100 mg, PO, once per day of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant. Participants also received gemcitabine, 1000 mg/m^2, IV, over 30 minutes on Days 1, 8 and 15 of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant.
Period: Overall Study
Arm/Group | Erlotinib, Gemcitabine: Rash Grade Less Than (<) 2 | Erlotinib, Gemcitabine: Rash Grade Greater Than/Equal to (≥) 2
Started | 115 | 38
Completed | 0 | 0
Not Completed | 115 | 38
Not completed — Adverse Event | 17 | 7
Not completed — Lack of Efficacy | 68 | 20
Not completed — Physician Decision | 10 | 4
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Other | 4 | 4
Not completed — Death | 8 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all participants included in the study.
Groups:
- Erlotinib, Gemcitabine: Rash Grade < 2: Participants with a rash Grade < 2 according to the National NCI-CTC V 3.0 received erlotinib, 100 mg, PO, once per day of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant. Participants also received gemcitabine, 1000 mg/m^2, IV, over 30 minutes on Days 1, 8 and 15 of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant.
- Erlotinib, Gemcitabine: Rash Grade ≥ 2: Participants with a rash Grade ≥ 2 according to the NCI-CTC V 3.0 received erlotinib, 100 mg, PO, once per day of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant. Participants also received gemcitabine, 1000 mg/m^2, IV, over 30 minutes on Days 1, 8 and 15 of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant.
- Total: Total of all reporting groups
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2 | Total
Number analyzed (Participants) | 115 | 38 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.9) | 62.0 (10.6) | 63.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 10 | 71
  Male | 54 | 28 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died During the Study
Time Frame: Enrollment through Cycle 24 (4-week cycles), up to 24 months.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 115 | 38
participants | 102 | 27

2. Primary Outcome: Overall Survival (OS) During the Study
Description: OS was defined as the time, in months, from the date of enrollment to the date of death due to any cause. Participants whose last recorded status was not death were censored. OS was estimated using Kaplan-Meier methodology.
Time Frame: Enrollment through Cycle 24 (4-week cycles), up to 24 months.
Population: ITT population; only participants who died were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 102 | 27
months | 4.468 [3.618 to 5.318] | 10.546 [9.679 to 11.414]

3. Secondary Outcome: Number of Participants Who Died at 6 Months
Time Frame: Enrollment through Cycle 6 (4-week cycles), up to 6 months.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 115 | 38
participants | 69 | 8

4. Secondary Outcome: OS At 6 Months
Description: as for outcome 2
Time Frame: Enrollment through Cycle 6 (4-week cycles), up to 6 months.
Population: ITT population; only participants who died were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 69 | 8
months | 4.468 [3.618 to 5.318] | NA [NA to NA] — The median and 95% confidence interval could not be calculated because of the large number of censored events.

5. Secondary Outcome: Number of Participants Who Died During the Study By Rash Grade
Time Frame: Enrollment through Cycle 24 (4-week cycles), up to 24 months.
Population: ITT population
Measure: Number; unit: participants
Groups:
- Erlotinib, Gemcitabine: Rash Grade 0: Participants with a rash Grade 0 according to the National NCI-CTC V 3.0 received erlotinib, 100 mg, PO, once per day of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant. Participants also received gemcitabine, 1000 mg/m^2, IV, over 30 minutes on Days 1, 8 and 15 of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant.
- Erlotinib, Gemcitabine: Rash Grade 1: Participants with a rash Grade 1 according to the National NCI-CTC V 3.0 received erlotinib, 100 mg, PO, once per day of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant. Participants also received gemcitabine, 1000 mg/m^2, IV, over 30 minutes on Days 1, 8 and 15 of Cycles 1 up through a maximum of Cycle 24 (4-week cycles) until disease progression, unacceptable toxicity, or treatment refusal by participant.
Arm/Group | Erlotinib, Gemcitabine: Rash Grade 0 | Erlotinib, Gemcitabine: Rash Grade 1 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 71 | 44 | 38
participants | 65 | 37 | 27

6. Secondary Outcome: OS By Rash Grade
Description: as for outcome 2
Time Frame: Enrollment through Cycle 24 (4-week cycles), up to 24 months.
Population: ITT population; only participants who died were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib, Gemcitabine: Rash Grade 0 | Erlotinib, Gemcitabine: Rash Grade 1 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 65 | 37 | 27
months | 3.318 [2.446 to 4.191] | 6.571 [5.139 to 8.003] | 10.546 [9.679 to 11.414]

7. Secondary Outcome: Number of Participants With Disease Progression or Death
Description: Progression-free survival (PFS) was defined as the time from the date of enrollment to the date of document disease progression or death due to any cause. As per Response Evaluation Criteria in Solid Tumors (RECIST) V 1.0, progressive disease (PD) was defined for target lesions (TLs) as at least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded since the start of treatment, and for non-target lesions (NTLs) as unequivocal progression of NTLs. Participants whose last recorded status was not PD or death were censored.
Time Frame: Enrollment, every 2 treatment cycles (4-week cycles) until disease progression, death, or end of study, for up to 24 months.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 115 | 38
participants | 110 | 33

8. Secondary Outcome: PFS
Description: The time, in months, from enrollment to PFS event. Participants whose last recorded status was not progression or death were censored. PFS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 7
Population: ITT population; only participants with an event (death or disease progression) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 110 | 33
months | 2.497 [2.130 to 2.864] | 6.439 [4.919 to 7.960]

9. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) According to RECIST
Description: As per RECIST V 1.0: for TLs, a CR was defined as the disappearance of all TLs; and a PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline (BL) SLD. For NTLs, a CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. Participants for whom no assessment of response was available and who had finalized the study due to disease progression or tumor-related death, disease progression was considered the BOR.
Time Frame: as for outcome 7
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 115 | 38
percentage of participants | 7.0 | 21.1
Statistical Analysis 1: Comparison: Erlotinib, Gemcitabine: Rash Grade < 2 vs Erlotinib, Gemcitabine: Rash Grade ≥ 2; Test type: Superiority or Other; p < 0.05, Chi-squared

10. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST
Description: Disease control was defined as BOR of CR, PR, or stable disease (SD). As per RECIST V 1.0: for TLs, a CR was defined as the disappearance of all TLs; and a PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the BL SLD; SD was defined as neither sufficient decrease in SLD to qualify for PR nor sufficient increase in SLD to qualify for PD. For NTLs, a CR was defined as the disappearance of all NTLs and normalization of tumor marker levels; SD was defined as the persistence of one or more NTLs and/or maintenance of tumor marker level above the normal limits. Participants for whom no assessment of response was available and who had finalized the study due to disease progression or tumor-related death, disease progression was considered the BOR.
Time Frame: as for outcome 7
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Number analyzed (Participants) | 115 | 38
percentage of participants | 42.6 | 84.2
Statistical Analysis 1: Comparison: Erlotinib, Gemcitabine: Rash Grade < 2 vs Erlotinib, Gemcitabine: Rash Grade ≥ 2; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded at every study visit for up to a maximum of 24 treatment cycles.
Description: All participants who received at least 1 dose of study treatment were included in the safety analysis.
Arm/Group | Erlotinib, Gemcitabine: Rash Grade < 2 | Erlotinib, Gemcitabine: Rash Grade ≥ 2
Serious Adverse Events (participants affected / at risk) | 58/115 | 14/38
Other Adverse Events (participants affected / at risk) | 115/115 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib, Gemcitabine: Rash Grade < 2 (N=115) | Erlotinib, Gemcitabine: Rash Grade ≥ 2 (N=38)
Haemorrhage, GI (Gastrointestinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Benign prostatic hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Sudden death (General disorders) | 1 | 0
Bilirubin (Hyperbilirubinemia) (Hepatobiliary disorders) | 1 | 0
Haemorrhage, rectal (Gastrointestinal disorders) | 1 | 0
Liver (Surgical and medical procedures) | 1 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Valvular heart disease (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 4 | 1
Fever (General disorders) | 4 | 2
Weight loss (Investigations) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal syndrome (Gastrointestinal disorders) | 1 | 0
Obstruction, GI (Gastrointestinal disorders) | 11 | 2
Perforation, GI (Gastrointestinal disorders) | 1 | 0
Visceral arterial ischemia (Gastrointestinal disorders) | 1 | 0
Haemorrhage, CNS (Nervous system disorders) | 1 | 0
Liver dysfunction (Hepatobiliary disorders) | 1 | 0
Liver dysfunction/failure (Hepatobiliary disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Anal/perianal (Infections and infestations) | 1 | 0
Blood (Infections and infestations) | 4 | 2
Cellulitis (Infections and infestations) | 1 | 0
Lung (pneumonia) (Infections and infestations) | 3 | 3
Peritoneal cavity (Infections and infestations) | 1 | 1
Upper airway nos (Infections and infestations) | 1 | 0
Urinary tract nos (Infections and infestations) | 1 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 0
CNS Cerebrovascular ischemia (Nervous system disorders) | 1 | 2
Confusion (Psychiatric disorders) | 1 | 0
Speech impairment (Nervous system disorders) | 0 | 1
Abdomen nos (Gastrointestinal disorders) | 5 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Obstruction, GU (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Thrombosis/Embolism (Vascular disorders) | 3 | 1
Thrombosis/Thrombus (Vascular disorders) | 3 | 0
Visceral arterial ischemia (Vascular disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Diabetes (Metabolism and nutrition disorders) | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib, Gemcitabine: Rash Grade < 2 (N=115) | Erlotinib, Gemcitabine: Rash Grade ≥ 2 (N=38)
Nausea (Gastrointestinal disorders) | 43 | 12
Constipation (Gastrointestinal disorders) | 38 | 12
Vomiting (Gastrointestinal disorders) | 34 | 8
Neutropenia (Blood and lymphatic system disorders) | 20 | 16
Anorexia (Metabolism and nutrition disorders) | 62 | 11
Weight loss (Investigations) | 27 | 5
Fever (General disorders) | 18 | 11
Fatigue (General disorders) | 89 | 31
Dysgeusia (Nervous system disorders) | 4 | 5
Ascites (Gastrointestinal disorders) | 7 | 2
Insomnia (Psychiatric disorders) | 4 | 2
Flatulence (Gastrointestinal disorders) | 3 | 2
Cataract (Eye disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Oral cavity (Gastrointestinal disorders) | 0 | 1
Esophagitis (Infections and infestations) | 1 | 1
Hypertension (Vascular disorders) | 2 | 1
Pulmonary hypertension (Vascular disorders) | 0 | 1
Myelitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1
Tremor (Nervous system disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Neuropathy (Nervous system disorders) | 6 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 0
Eyelid dysfunction (Eye disorders) | 1 | 0
Ocular surface disease (Eye disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Monocytopenia (Blood and lymphatic system disorders) | 1 | 0
Proctitis (Infections and infestations) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Vision - Blurred vision (Eye disorders) | 1 | 0
Allergy /immunology- other (Immune system disorders) | 2 | 0
Hearing loss (Ear and labyrinth disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 32 | 11
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 3 | 1
Hemorrhage (Blood and lymphatic system disorders) | 1 | 0
Leukocytes (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 8 | 3
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Constitutional symptoms- other (General disorders) | 11 | 6
Sweating (Metabolism and nutrition disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Cheilitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatology/skin- other (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 1
Diabetes (Metabolism and nutrition disorders) | 2 | 1
Endocrine- other (Endocrine disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 55 | 15
Gastrointestinal - other (Gastrointestinal disorders) | 21 | 5
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 13 | 3
Hemorrhoids (Gastrointestinal disorders) | 3 | 1
Mucositis/stomatitis (Gastrointestinal disorders) | 19 | 9
Obstruction, GI (Gastrointestinal disorders) | 2 | 1
Perforation, GI (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Xerostomia (Gastrointestinal disorders) | 6 | 2
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hemorrhage rectal (Gastrointestinal disorders) | 1 | 0
Liver dysfunction (Hepatobiliary disorders) | 8 | 3
Pancreas, exocrine (Gastrointestinal disorders) | 3 | 0
Abdomen nos (Infections and infestations) | 0 | 1
Anal/perianal (Infections and infestations) | 1 | 0
Blood (Infections and infestations) | 1 | 1
Conjunctiva (Infections and infestations) | 5 | 0
Infection (Infections and infestations) | 1 | 0
Lung (Pneumonia) (Infections and infestations) | 1 | 1
Middle ear (Infections and infestations) | 0 | 1
Oral cavity-gums (Infections and infestations) | 2 | 0
Skin (Infections and infestations) | 3 | 0
Soft tissue nos (Infections and infestations) | 1 | 0
Upper airway nos (Infections and infestations) | 6 | 3
Urinary tract nos (Infections and infestations) | 3 | 1
Edema (Blood and lymphatic system disorders) | 11 | 3
Edema: limb (Blood and lymphatic system disorders) | 22 | 2
Lymphatics- other (Blood and lymphatic system disorders) | 1 | 0
Albumin, serum-low (Metabolism and nutrition disorders) | 1 | 0
Alkaline phosphatase (Investigations) | 3 | 0
ALT, SGPT (Investigations) | 1 | 1
ALT, SGPT (Investigations) | 4 | 2
Bilirubin (Hepatobiliary disorders) | 4 | 4
Calcium, serum high (Metabolism and nutrition disorders) | 4 | 1
GGT (Gamma-glutamyl) (Investigations) | 5 | 1
Glucose, serum high (Metabolism and nutrition disorders) | 6 | 1
Glucose, serum low (Metabolism and nutrition disorders) | 5 | 1
Hypercreatinaemia (Metabolism and nutrition disorders) | 0 | 1
Magnesium, serum low (Metabolism and nutrition disorders) | 3 | 1
Metabolic/laboratory (Metabolism and nutrition disorders) | 3 | 1
Potassium, serum high (Metabolism and nutrition disorders) | 1 | 1
Potassium, serum low (Metabolism and nutrition disorders) | 3 | 0
Dizziness (Nervous system disorders) | 3 | 2
Extrapyramidal (Nervous system disorders) | 0 | 1
Personality/behavioral (Psychiatric disorders) | 19 | 2
Somnolence (Nervous system disorders) | 4 | 0
Other (General disorders) | 1 | 0
Abdomen nos (Musculoskeletal and connective tissue disorders) | 78 | 19
Back (Musculoskeletal and connective tissue disorders) | 9 | 7
Bone (Musculoskeletal and connective tissue disorders) | 4 | 0
Chest/thorax nos (General disorders) | 2 | 0
Genitourinary (Renal and urinary disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 1
Joint (Musculoskeletal and connective tissue disorders) | 2 | 0
Kidney (Renal and urinary disorders) | 1 | 0
Muscle (Musculoskeletal and connective tissue disorders) | 5 | 6
Neck (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck/back (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain (General disorders) | 18 | 8
Peritoneum (General disorders) | 1 | 0
Skin (General disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Nasal/ paranasal (General disorders) | 1 | 1
Nasal/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonay/upper respiratoy- other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cystitis (Infections and infestations) | 6 | 2
Incontinence, urinary (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 1
Renal/genitourinary (Renal and urinary disorders) | 1 | 0
Testicular oedema (Reproductive system and breast disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Urine color change (Renal and urinary disorders) | 6 | 0
Upper airway nos (Surgical and medical procedures) | 1 | 0
Vein nos (Surgical and medical procedures) | 1 | 0
Phlebitis (Vascular disorders) | 5 | 4
Thrombosis/embolism (Vascular disorders) | 7 | 5
Thrombosis/thrombus (Vascular disorders) | 4 | 0
Vein injury (Vascular disorders) | 0 | 1
Distension/bloating (Gastrointestinal disorders) | 3 | 3
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Ocular/visual- other (Eye disorders) | 2 | 0
Thrombopenia (Blood and lymphatic system disorders) | 21 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.